CLINICAL TRIAL: NCT00502983
Title: Molecular Epidemiology of Acute Myelogenous Leukemia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ID03-0250
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Leukemia
Keywords: Acute Myelogenous Leukemia; Epidemiology; Leukemia; Healthy Control; Lifestyle Factors; Genetic Susceptibility; Interview; AML
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Genetic Predisposition to Disease | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample collection to look for any biologic factors associated with AML.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Interview: AML Patients & Healthy Controls
  Interventions: Behavioral: Interview

INTERVENTIONS:
Behavioral: Interview — Interview lasting approximately 50 minutes.

SUMMARY:
Little is known about the epidemiologic risk factors associated with the development of acute myelogenous leukemia (AML), and less is known about the role that genetic susceptibility plays in the development of AML. We propose to conduct a population-based study to investigate genetic susceptibility in adult AML patients, both de novo and treatment-related in a well-defined geographical area. Using a case-control design, we will prospectively enroll 400 patients from Texas and 800 healthy controls. Controls will be recruited using random digit dialing, and will be matched to the cases by age, gender, and ethnicity. Epidemiological and demographic information will be obtained through personal interviews, and will be integrated with clinical information, cytogenetic data, and genotypic markers. Blood specimens will be collected on all participants, who will be genotyped for markers associated with activation and detoxification of chemical carcinogens, including chemotherapy drugs. Polymorphisms in genes such as cytochrome p450 (CYP2E1), glutathione S-transferases (GSTT1, GSTM1, GSTP1), epoxide hydrolase (HYL1), NADPH-quinone oxidoreductase (NQO1), and myeloperoxidase (MPO) will be analyzed.

This study will provide insight into the role that these susceptibility markers, along with clinical epidemiological, and cytogenetic factors, play in the identification of people at risk of developing AML. Understanding how genetic predisposition and exogenous exposures interact to determine AML susceptibility will allow the development of prevention strategies in the future.

DETAILED DESCRIPTION:
INFORMED CONSENTS FOR AML PATIENTS:

For this study, participant will be asked to complete a personal interview. During the interview, participant will be asked questions about participant's demographics (age, sex, etc.), any chemicals participant may have been exposed to, participant's medical history, family history of cancer, participant's diet, and participant's smoking and alcohol use histories. It should take around 50 minutes to complete the interview.

Participant will also have around 1 tablespoon of blood drawn for special tests. These tests will look for any biologic factors associated with AML.

The interview and the blood draw may be done during a regularly scheduled visit to M. D. Anderson, or may be scheduled at the time and place of participant's convenience.

Participant may be contacted at home by phone so that researchers can collect information about any changes in participant's health status.

This is an investigational study. Up to 1,200 participants will take part in this study.

INFORMED CONSENT FOR CONTROL SUBJECTS:

For this study, participant will be asked to complete a personal interview. During the interview, participant will be asked questions about participant's demographics (age, sex, etc.), any chemicals participant may have been exposed to, participant's medical history, family history of cancer, participant's diet, and participant's smoking and alcohol use histories. It should take around 50 minutes to complete the interview.

Participant will also have around 1 tablespoon of blood drawn for special tests. These tests will look for any biologic factors associated with AML. The interview and blood draw will be scheduled at the time and place of participant's convenience.

This is an investigational study. Up to 1,200 participants will take part in this study.

ELIGIBILITY:
Inclusion Criteria:

1. A histologically confirmed diagnosis of AML (patients only)
2. Aged 18 or older
3. Resident of Texas
4. Willing and able to provide written informed consent and authorization
5. Willing to donate 10mL of blood and complete a personal interview

Exclusion Criteria:

1. Under 18 years of age
2. History of invasive cancer, excluding non-melanoma skin cancer (controls only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: UT MDACC Patients with Acute Myelogenous Leukemia and healthy controls, all 18 years of age or older and Texas residents.
Sampling Method: Non-Probability Sample
Enrollment: 519 (Actual)
Dates: Start 2003-06-23 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Identify biologic and lifestyle factors that may increase a person's risk of developing acute myelogenous leukemia. | 8 Years

CONTACTS AND LOCATIONS:
Overall Officials: Jian Gu, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org